CLINICAL TRIAL: NCT00423579
Title: A Multicenter, Randomized, Parallel-Groups, Double-Blind Placebo-Controlled Study Comparing the Efficacy, Safety, and Tolerability of Administration of Ezetimibe/Simvastatin Tablet 10/20 mg Versus Doubling the Dose of Simvastatin 20 mg [Simvastatin 40 mg] in Subjects With Primary Hypercholesterolemia and Coronary Heart Disease
Brief Title: The Effects of Ezetimibe/Simvastatin 10/20 mg Versus Simvastatin 40 mg in High Cholesterol and Coronary Heart Disease Study (P04039AM2)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P04039
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Results first posted 2009-08-25 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Coronary Disease
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease | interventions — Ezetimibe; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ezetimibe/Simvastatin 10/20 mg + Simvastatin placebo (Experimental): Subjects will receive 2 tablets. The first tablet is Ezetimibe/Simvastatin 10/20 mg. The second tablet is simvastatin placebo. Subjects will receive a maximum of 6 weeks of treatment
  Interventions: Drug: Ezetimibe/Simvastatin 10/20 mg
- Ezetimibe/Simvastatin placebo + Simvastatin 40 mg (Active Comparator): Subjects will receive 2 tablets. The first tablet is Ezetimibe/Simvastatin placebo. The second tablet is simvastatin 40 mg. Subjects will receive a maximum of 6 weeks of treatment.
  Interventions: Drug: simvastatin 40 mg

INTERVENTIONS:
Drug: Ezetimibe/Simvastatin 10/20 mg — 1 tablet containing 10 mg of ezetimibe and 20 mg of simvastatin per day for 6 weeks
  Arms: Ezetimibe/Simvastatin 10/20 mg + Simvastatin placebo
Drug: simvastatin 40 mg — 1 tablet containing 40 mg of simvastatin per day for 6 weeks
  Arms: Ezetimibe/Simvastatin placebo + Simvastatin 40 mg

SUMMARY:
This study is being conducted to compare the efficacy, safety, and tolerability of ezetimibe/simvastatin 10/20 mg when administered daily versus doubling the dose of simvastatin to 40 mg in patients with hypercholesterolemia and coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have documented coronary heart disease (CHD). For the purposes of this study, CHD will include one or more of the following features: documented stable angina (with evidence of ischemia on exercise testing); history of myocardial infarction; history of percutaneous coronary intervention [PCI] (primarily PCI with or without stent placement); symptomatic peripheral vascular disease (claudication); documented history of atherothrombotic cerebrovascular disease; and/or documented history of unstable angina or non-Q wave myocardial infarction.
* Subjects must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* History of myocardial infarction (heart attack).
* Subjects must be >= 18 years and <= 75 years of age.
* Subjects must have an LDL-C concentration >= 2.6 mmol/L (100 mg/dL) to <= 4.1 mmol/L (160 mg/dL) at the time of randomization (Visit 3/Baseline Visit).
* Subjects must have triglyceride concentrations of < 3.99 mmol/L (350 mg/dL) at (Visit 3 Baseline Visit).
* Subject must be currently taking simvastatin 20 mg daily.
* Subjects must have liver transaminases (ALT [alanine aminotransferase], AST [aspartate aminotransferase]) < 50% above the upper limit of normal, with no active liver disease, and CK (creatine kinase) < 50% above the upper limit of normal at Visit 3 (Baseline Visit).
* Clinical laboratory tests (complete blood count [CBC], blood chemistries, urinalysis) must be within normal limits or clinically acceptable to the investigator at Visit 3 (Baseline Visit).
* Subjects must have maintained a cholesterol-lowering diet and exercise program for at least 4 weeks prior to the study and be willing to continue the same diet and exercise program during the study.
* Subjects must report a stable weight history for at least 4 weeks prior to entry into study at Visit 3 (Baseline Visit).
* Women receiving hormonal therapy, including hormone replacement, any estrogen antagonist/agonist, or oral contraceptives, must have been maintained on a stable dose and regimen for at least 8 weeks and be willing to continue the same regimen for the duration of the study.
* Women of childbearing potential (includes women who are less than 1 year postmenopausal and women who become sexually active) must be using an acceptable method of birth control (e.g., hormonal contraceptive, medically prescribed intrauterine device [IUD], condom in combination with spermicide) or be surgically sterilized (e.g., hysterectomy or tubal ligation).
* Subjects must be free of any clinically significant diseases other than hyperlipidemia or coronary heart disease that would interfere with study evaluations.
* Subjects must understand and be able to adhere to the dosing and visit schedules, and must agree to remain on their cholesterol-lowering diet and their exercise regimen for the duration of the study.

Exclusion Criteria:

* Subjects whose body mass index (BMI = weight [kg]/height2 [m]) is >= 35 kg/m^2 at Visit 3 (Baseline Visit).
* Subjects who consume > 14 alcoholic drinks per week. (A drink is: a can of beer, glass of wine, or single measure of spirits).
* Any condition or situation which, in the opinion of the investigator, might pose a risk to the subject or interfere with participation in the study.
* Women who are pregnant or nursing.

Exclusion Criteria: subjects who have the following medical conditions:

* Congestive heart failure defined by New York Heart Association (NYHA) as Class III or IV.
* Uncontrolled cardiac arrhythmia.
* Myocardial infarction, acute coronary insufficiency, coronary artery bypass surgery, or angioplasty within 3 months of Visit 3 (Baseline Visit).
* Unstable or severe peripheral artery disease within 3 months of Visit 3 (Baseline Visit).
* Newly diagnosed or currently unstable angina pectoris (chest pain).
* Uncontrolled hypertension (treated or untreated) with systolic blood pressure > 160 mm Hg or diastolic > 100 mm Hg at Visit 3 (Baseline Visit).
* Type I or Type II diabetes mellitus.
* Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins, i.e., secondary causes of hyperlipidemia, such as secondary hypercholesterolemia due to hypothyroidism (thyroid stimulating hormone [TSH] above upper limit of normal) at Visit 3. Subjects with a history of hypothyroidism who are on a stable therapy of thyroid hormone replacement for at least 6 weeks are eligible for enrollment if TSH levels are within normal limits at Visit 3 (Baseline Visit).
* Impaired renal function (creatinine > 2.0 mg/dL) or nephrotic syndrome at Visit 3 (Baseline Visit).
* Disorders of the hematologic, digestive, or central nervous systems including cerebrovascular disease and degenerative disease that would limit study evaluation or participation.
* Known Human Immunodeficiency Virus (HIV) positive.
* Cancer within the past 5 years (except for successfully treated basal and squamous cell carcinomas).
* History of mental instability, drug/alcohol abuse within the past 5 years, or major psychiatric illness not adequately controlled and stable on pharmacotherapy.

Exclusion Criteria: subjects who are on any of the following concomitant medications:

* Subjects who have not observed the designated wash-out period for any of the prohibited medications.
* Subjects who have not stopped taking various prohibited medications for a minimum period of time before Visit 3, including amiodarone hydrochloride (6 months) and probucol (12 months).
* Subjects currently consuming large amounts of grapefruit juice (> 1 liter/day).
* Oral corticosteroids, unless used as replacement therapy for pituitary/adrenal disease and the subject is on a stable regimen for at least 6 weeks prior to Visit 3 (Baseline Visit).
* Subjects who are currently using cardiovascular medication (e.g. antihypertensive, antiarrhythmic) and have not been on a stable regimen for at least 6 weeks prior to Visit 3 (Baseline Visit) and it is expected to change during the study.
* Subjects who are currently using psyllium, other fiber-based laxatives, and/or any other over-the-counter (OTC) therapy known to affect serum lipid levels (phytosterol margarine), and have not been on a stable regimen for at least 5 weeks prior to study entry Visit 3 (Baseline Visit) and who do not agree to remain on this regimen throughout the study.
* Subject who are currently using orlistat or sibutramine.
* Subjects who are currently using amiodarone hydrochloride.
* Subjects who are currently using danazol.
* Subjects who are currently using coumarin anticoagulants (warfarin).
* Subjects who are using (at the Screening Visit / Visit 1) any statin other than simvastatin 20 mg, or ezetimibe alone or in combination with any statin (including the fixed combination with simvastatin).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-07-01 (Actual); Primary Completion 2008-03-01 (Actual); Study Completion 2008-03-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Averna M, Zaninelli A, Le Grazie C, Gensini GF. Ezetimibe/simvastatin 10/20 mg versus simvastatin 40 mg in coronary heart disease patients. J Clin Lipidol. 2010 Jul-Aug;4(4):272-8. doi: 10.1016/j.jacl.2010.05.002. Epub 2010 Jun 1. PMID 21122660
- [Derived] Rotella CM, Zaninelli A, Le Grazie C, Hanson ME, Gensini GF. Ezetimibe/simvastatin vs simvastatin in coronary heart disease patients with or without diabetes. Lipids Health Dis. 2010 Jul 27;9:80. doi: 10.1186/1476-511X-9-80. PMID 20663203

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Visits 1 and 2 were for screening, combined if wash-out not required. One ineligible subject mistakenly received assignment at Visit 2 and was removed. The subject did not receive treatment. Actual enrollment: 120 subjects. Intent-to-treat (ITT) population included only evaluable subjects; as such analysis based on 112 subjects.
Groups:
- Ezetimibe/Simvastatin 10/20 mg + Simvastatin Placebo: Subjects in the Intent-to-Treat Population. Subjects will receive 2 tablets. The first tablet is Ezetimibe/Simvastatin 10/20 mg. The second tablet is simvastatin placebo. Subjects will receive a maximum of 6 weeks of treatment
- Ezetimibe/Simvastatin Placebo + Simvastatin 40 mg: Subjects in the Intent-to-Treat population. Subjects will receive 2 tablets. The first tablet is Ezetimibe/Simvastatin placebo. The second tablet is simvastatin 40 mg. Subjects will receive a maximum of 6 weeks of treatment.
Period: Overall Study
Arm/Group | Ezetimibe/Simvastatin 10/20 mg + Simvastatin Placebo | Ezetimibe/Simvastatin Placebo + Simvastatin 40 mg
Started | 60 (61 enrolled, however one subject was ineligible and was removed.) | 60
Completed | 56 (These 56 subjects were the Intent-to-Treat population. Analysis based on ITT population.) | 56 (These 56 subjects were the Intent-to-Treat population. Analysis based on ITT population.)
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 3 | 0
Not completed — Protocol Violation | 1 | 3
Not completed — Diagnosis of diabetes | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe/Simvastatin 10/20 mg + Simvastatin Placebo | Ezetimibe/Simvastatin Placebo + Simvastatin 40 mg | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age based on Intent-to-Treat population.
  years | 61.3 (8.4) | 62.1 (7.8) | 61.7 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender totals based on Intent-to-Treat population.
  Participants
    Female | 26 | 24 | 50
    Male | 30 | 32 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change in Low-density-lipoprotein Cholesterol (LDL-C) at 6 Weeks
Description: Percentage change in LDL C from baseline to endpoint after 6 weeks of treatment.
Time Frame: Baseline and 6 weeks
Population: Intent-to-treat population only.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Ezetimibe/Simvastatin 10/20 mg + Simvastatin Placebo | Ezetimibe/Simvastatin Placebo + Simvastatin 40 mg
Number analyzed (Participants) | 56 | 56
percentage change | -26.5 (9.5) | -11.9 (13.6)
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin 10/20 mg + Simvastatin Placebo vs Ezetimibe/Simvastatin Placebo + Simvastatin 40 mg; Test type: Superiority or Other; p = 0.0000, Student's t test for independent data; Mean Difference (Net) = -14.5, 95% CI [-18.9 to -10.1] — Difference in percentage change in mean LDL-C values (change from baseline to week 6) between the two treatment groups. (Ezetimibe [EZ]/Simvastatin [S] [10/20mg] + S [placebo] group minus the EZ/S [10mg/placebo] + S [40mg] group)

ADVERSE EVENTS:
Arm/Group | Ezetimibe/Simvastatin 10/20 mg + Simvastatin Placebo | Ezetimibe/Simvastatin Placebo + Simvastatin 40 mg
Serious Adverse Events (participants affected / at risk) | 0/60 | 1/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe/Simvastatin 10/20 mg + Simvastatin Placebo (N=60) | Ezetimibe/Simvastatin Placebo + Simvastatin 40 mg (N=60)
Transient Ischemic Attack (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall not publish or publicly present the study results without prior written authorization from the sponsor, except for dispositions in the Ministerial Circular n. 6 dated 02 SEP 2002. The investigator shall notify the sponsor in writing of any publication submission or presentation reporting results of the study 30 days prior to submission or presentation to permit sponsor review.